CLINICAL TRIAL: NCT03832543
Title: Modified Extraperitoneal Uterosacral Ligament Suspension in Preventing Cuff Prolapse Risk After Vaginal Hysterectomy; 4 Clamp Method
Brief Title: Modified Uterosacral Ligament Suspension in Vaginal Hysterectomy
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kerem Doga Seckin, Ass. Prof Kerem Doga Seckin, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 0651603
Record Dates: First submitted 2019-02-02; First posted 2019-02-06 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Modified Extraperitoneal Uterosacral Ligament Suspension; Vault Prolapse, Vaginal
Keywords: Vaginal Hysterectomy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction : The extraperitoneal uterosacral ligament suspension (ULS) can be performed during the removal of the uterus in vaginal hysterectomy to prevent cuff prolapse. In this study, the modified extraperitoneal ULS technique was evaluated in terms of preventing cuff prolapse.

Methods / Technique : Forty patients with second and third-stage uterine prolapse who were operated were included in the study. During routine vaginal hysterectomy procedure performed on patients, after sacrouterine ligaments which are the first-bites and uteroovarian and round ligaments which are the last-bites have been sutured and knotted, these ligaments were marked with 4-distinct clemps to make the right and left, upper and lower separation. After vaginal cuff was closed the sutures hanged by the clamps were ligated together, and the cuff tissue was stretched to the apical line.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2 or 3 uterin prolapse

Exclusion Criteria:

* contrandication for surgery

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 40-75 years old
Study Population: Stage 2 or 3 uterin prolapse who need surgery
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
postoperative vaginal cuff prolapse | 2 years
  During two years follow up after sugery if there is vaginal cuff prolapse or not. The measurement of the vaginal cuff distance to the hymenal ring with a calculator. The units were centimeter

IPD SHARING:
Plan to Share IPD: No